CLINICAL TRIAL: NCT06573476
Title: Addressing Racial Disparities in Opioid Overdose Deaths Using an Open Source Peer Recovery Coach Training and Multimodal Mobile Health Platform
Brief Title: Addressing Racial Disparities in Opioid Overdose Using Peer Recovery Coach Training and mHealth Platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA059770 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; Peer Recovery Coach; Cultural Structural Humility; mHealth; People With Opioid Use Disorder; OUD; PWOUD; mHealth Intervention
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Arm-1: PRC supported text+ AI driven CSDH-enhanced text (Experimental): Individuals randomized to Arm-1 will receive PRC-supported text check-ins and AI-driven CSDH-enhanced text messaging.
  Interventions: Behavioral: PRC supported text + AI driven CSDH-enhanced text
- Intervention Arm-2: AI driven CSDH-enhanced text only (Experimental): Individuals randomized to Arm-2 will receive the AI-driven CSDH-enhanced text messaging only
  Interventions: Behavioral: AI driven CSDH-enhanced text only
- Control Arm 3- Treatment as Usual (Placebo Comparator): Individuals randomized to the control arm will receive treatment as usual.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: PRC supported text + AI driven CSDH-enhanced text — In interventional Arm-1, PRC-supported text check-ins to participants (3x/week) will be provided by PRC study staff in addition to automated AI-driven texts. The PRC will personalize text "check-ins" to participants based on: (a) baseline CSDH needs (e.g., food insecurity, legal aid); (b) initial intake visit in primary care or challenges with service entry; and (c) content outlined in the CSH training addressing emerging participant challenges.
  Arms: Intervention Arm-1: PRC supported text+ AI driven CSDH-enhanced text
Behavioral: AI driven CSDH-enhanced text only — In interventional Arm-2, participants will receive the AI-driven CSDH-enhanced text messaging only. Participants in this arm will not receive text support from the PRC.
  Arms: Intervention Arm-2: AI driven CSDH-enhanced text only
Behavioral: Treatment as Usual (TAU) — In Arm-3, the control group, individuals randomized to the control arm will receive treatment as usual (i.e., verbal instructions and NYC Dept of Health pamphlets detailing access to OUD and social services). No services will be provided except for social/clinical service referrals given at the end of each REDCap visit.
  Arms: Control Arm 3- Treatment as Usual

SUMMARY:
The study aims to adapt an existing Cultural Structural Humility (CSH) training into a video format for peer recovery coaches (PRCs) and refine an AI-driven texting tool to reinforce the training. After refining these tools using user-centered design, a pilot test will be conducted to assess their impact on the uptake of opioid treatment and social services. The study will also evaluate the feasibility and effectiveness of the intervention to inform future large-scale trials.

DETAILED DESCRIPTION:
The purpose of this study is to adapt an evidence-supported, currently staff-led Cultural Structural Humility (CSH) training to an interactive video format (7 brief video modules) for PRCs (Aim 1) while concurrently, refining a validated AI-driven texting tool that will newly reinforce core CSH training principles (Aim 2) that focus upon cultural and structural determinants of health (CSDH). After completing iterative refinement per user-centered design strategies based on the Technology Acceptance Model (TAM) for Aim 1 and 2, the investigators will pilot test CSH-trained PRCs delivering telephone based care/services coordination combined with refined AI-driven texting to enhance uptake of MOUD services, and social services (Aim 3). Aim 3 is sized for feasibility testing, final 'de-bugging' of the platform, and informing study conceptualization for a future large-scale efficacy trial. In this R34, the intervention effects will be assessed on the primary clinical outcome (i.e., receipt of buprenorphine), secondary outcome (i.e., uptake of social services), and implementation of the proposed multimodal intervention platform per the RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* fluent in English
* self-reported non-prescription opioid use <30 days prior to consent
* provision of informed consent
* planned stay in NYC ≥3 months
* Black and/or Latinx race/ethnicity
* positive urine toxicology for opioids per EMR records or study staff administered random saliva drug testing
* diagnosis of OUD per the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
* self-reported interest in initiating buprenorphine in primary care, or elsewhere.

Exclusion Criteria:

* inability to comprehend text content written at a 3rd grade reading level
* physical or visual disability preventing mobile phone use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Estimated Rate of PRC-PWUO Contact | 3 months
  The number of contacts between Peer Recovery Coaches (PRC) and People Who Use Opioids (PWUO), measured through communication logs.
Rate of AI-Driven Texting Use Among PWUO | 3 months
  The frequency of AI-driven text interactions initiated by PWUO, captured through software logs.
Change in Felt and/or Anticipated Stigma | 3 months
  The change in felt and/or anticipated stigma pre- and post-intervention, measured by a validated stigma assessment questionnaire.
Amount of time to Initial Receipt of Buprenorphine (Self-Reported) | 3 months
  The time (in days) to the initial receipt of buprenorphine, as self-reported by participants.
The Amount of Self-Reported Social Services Use | 3 months
  The self-reported utilization of social services at baseline, 1 month, and 3 months, addressing social determinants of health (SDH) to assess intervention effect sizes.
Cost (Amount of Money) of Implementing and Sustaining the Multimodal Intervention | 3 months
  The associated cost of implementing and sustaining the multimodal intervention, including cost-per quality-adjusted life year (QALY) and cost-per opioid use disorder (OUD) treatment days.

SECONDARY OUTCOMES:
The Amount of Participants That Retain in Treatment | 3 months
  The number of participants continuously retained in buprenorphine treatment over a 12-week period, assessed at the 12-week mark.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ventuneac, Study Director — START Treatment and Recovery
Locations (1):
- START Treatment and Recovery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No